CLINICAL TRIAL: NCT07193810
Title: Exploratory Clinical Study on the Safety and Preliminary Efficacy of CC312 in the Treatment of Relapsed/Refractory Autoimmune Diseases
Brief Title: A Study of CC312 for Relapsed/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: CytoCares Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC312-I-003
Record Dates: First submitted 2025-09-15; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: SLE - Systemic Lupus Erythematosus; IIM- Idiopathic Inflammatory Myopathies; SSc-Systemic Sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CC312 (Experimental)
  Interventions: Biological: CC312

INTERVENTIONS:
Biological: CC312 — CC312 is administered twice weekly (BIW) on Day 1 and Day 4 of each week for a 4-week treatment period. After Day 28, subsequent dosing (including the decision to continue treatment, dosing frequency, and treatment duration) will be determined based on the subject's clinical response and B-cell depletion status. The maximum planned treatment period is 24 weeks, followed by a follow-up phase.

SUMMARY:
This study is an open-label, multiple ascending dose investigator-initiated trial (IIT) designed to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of CC312 in adult patients with relapsed or refractory autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the trial's purpose, nature, methodology, and potential adverse reactions, voluntarily participate as a subject, and sign the informed consent form.
* Aged 18-65 years (inclusive, based on the date of signing the informed consent form), regardless of gender.
* For Systemic Lupus Erythematosus (SLE):

  1. Diagnosed with SLE according to the 2019 EULAR/ACR classification criteria；
  2. Meet at least one of the following: positive antinuclear antibody (ANA) and/or anti-dsDNA antibody and/or anti-Sm antibody at screening；
  3. Had an inadequate response or relapse after standard therapy, defined as any of the following (alone or combined): glucocorticoids, antimalarials (hydroxychloroquine), immunosuppressants (including mycophenolate mofetil, cyclophosphamide, leflunomide, methotrexate, tacrolimus, cyclosporine, azathioprine), or biologics (rituximab, belimumab, telitacicept). Each regimen must have been administered for ≥3 months, and the subject must have received ≥2 immunosuppressants and/or biologics；
  4. At screening, meet SLEDAI-2000 ≥7 and have at least one BILAG A or two BILAG B organ domain scores；
  5. Prior to the first dose, subjects must have received glucocorticoids and/or antimalarials and/or immunosuppressants for ≥12 weeks, with stable doses for ≥30 days；
  6. If receiving oral glucocorticoids (e.g., prednisone), the dose must be ≤40 mg/day at screening and during the screening period；
  7. If using glucocorticoids alone, the dose must be ≥7.5 mg/day prednisone (or equivalent).
* For Idiopathic Inflammatory Myopathy (IIM):

  1. Diagnosed with possible or definite IIM per the 2017 EULAR/ACR classification criteria (≥5.5 points without biopsy; ≥6.7 points with biopsy) ；
  2. Have at least one positive myositis-specific autoantibody (MSA) , myositis-associated autoantibody (MAA), or ANA at or prior to screening；
  3. Had an inadequate response or relapse after conventional therapy, defined as glucocorticoids (prednisone >1 mg/kg/day or equivalent) and ≥1 immunomodulatory drug (immunosuppressants: azathioprine, mycophenolate mofetil, cyclophosphamide, methotrexate, leflunomide, tacrolimus, cyclosporine; biologics: rituximab, belimumab; small molecules: tofacitinib), each for ≥3 months, with ≥2 immunosuppressants and/or biologics used；
  4. Have active IIM at screening, defined as meeting ≥3 of MMT-8 total score ≤141/150 with ≥20% strength loss in affected muscles; Physician global activity ≥2; Patient global activity ≥2; MDAAT ≥2; ≥2 muscle enzymes elevated, with one ≥1.5× ULN; HAQ ≥0.25；
  5. Prior to the first dose, subjects must have received glucocorticoids and/or immunosuppressants for ≥12 weeks, with stable glucocorticoid doses for ≥30 days and immunosuppressant doses for ≥60 days. Glucocorticoid dose must be ≤60 mg/day prednisone during screening；
  6. If using glucocorticoids alone, the dose must be ≥7.5 mg/day prednisone.
* For Systemic Sclerosis (SSc):

  1. Diagnosed with diffuse cutaneous SSc per the 2013 EULAR/ACR criteria ；
  2. Have positive ANA and/or SSc-related antibodies (e.g., Scl70, Th/To, RP11/12, U3RNP)；
  3. Disease duration ≤5 years (from initial diagnosis)；
  4. Had an inadequate response or relapse after conventional therapy (glucocorticoids + ≥1 immunomodulator: cyclophosphamide, mycophenolate mofetil, methotrexate, leflunomide, azathioprine, tacrolimus, cyclosporine, and/or biologics), each for >6 months；
  5. mRSS ≥15 and ≤30 at screening with progression within 6 months；
  6. Prior to the first dose, subjects must have received glucocorticoids and/or immunosuppressants for ≥12 weeks, with stable glucocorticoid doses for ≥30 days and immunosuppressant doses for ≥60 days. Glucocorticoid dose must be ≤10 mg/day during screening.
* Females of childbearing potential must use highly effective contraception from screening until 6 months after the last dose, refrain from oocyte donation, and ensure male partners use effective contraception.
* Males of childbearing potential must use effective contraception from screening until 6 months after the last dose, with no plans for fertility or sperm donation, and ensure female partners use effective contraception.

Exclusion Criteria:

* Severe lupus nephritis within 8 weeks prior to screening (defined as urinary protein >6 g/24 h, serum creatinine >2.5 mg/dL or 221 μmol/L), requirement of prohibited medications for active nephritis per protocol, need for hemodialysis, or receipt of prednisone ≥100 mg/day (or equivalent glucocorticoids) for ≥14 days.
* Central nervous system disorders (including but not limited to epilepsy, psychosis, interstitial encephalopathy syndrome, cerebrovascular accident, encephalitis, or CNS vasculitis) within 8 weeks prior to screening.
* Other types of idiopathic inflammatory myopathies: inclusion body myositis, amyotrophic diabetes, or juvenile myositis; patients with severe muscle damage or permanent weakness/cardiac involvement due to non-IIM causes (e.g., stroke).
* SSc-related pulmonary hypertension requiring treatment; rapidly progressive SSc-related lower gastrointestinal (small/large intestine) involvement requiring parenteral nutrition; active gastric antral vascular ectasia; history of SSc-related renal crisis.
* History of major organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
* Other concurrent autoimmune diseases requiring systemic therapy.
* IgA deficiency (serum IgA level <10 mg/dL).
* Abnormal laboratory findings at screening: Liver function: AST/ALT >2× upper limit of normal (ULN) (except for IIM patients with elevated muscle enzymes); Hematology: hemoglobin <85 g/L, white blood cell count <2.5×10⁹/L, platelet count <50×10⁹/L.
* Participation in any other clinical trial (including cell or gene therapy) within 4 weeks prior to screening or within 5 half-lives of the investigational product (whichever is longer).
* Received CAR-T therapy within 6 months prior to screening.
* Treatment with B-cell-depleting agents (e.g., rituximab, or therapies targeting CD19/CD20/BAFF) within 1 month prior to screening, unless B-cell levels returned to pre-treatment or normal ranges.
* Received non-standard anti-SLE therapies (e.g., anifrolumab) within 3 months or 5 half-lives of the drug (whichever is longer) prior to screening.
* Received live/attenuated vaccination within 4 weeks prior to screening or plans to receive such during the trial.
* Active severe infection requiring antibiotic treatment within 14 days prior to screening.
* History of Grade 3-4 allergic reaction (per CTCAE v5.0) to another monoclonal antibody, or known hypersensitivity to any component of CC312 (e.g., recombinant proteins, polysorbate 80). Patients with transient (≤24 h) Grade ≤3 reactions may be included after discussion with the investigator.
* Evidence of drug abuse, substance abuse, or alcohol addiction.
* Major surgery within 4 weeks or minor surgery within 2 weeks prior to screening; wounds must be fully healed (procedures like catheter placement are excluded).
* History of cardiovascular events within 6 months prior to screening: NYHA Class III/IV heart failure, myocardial infarction, unstable angina, uncontrolled/symptomatic atrial arrhythmia, ventricular arrhythmia, or other clinically significant cardiac conditions.
* Any other severe underlying disease (e.g., active gastric ulcer, uncontrolled seizures, cerebrovascular events, GI bleeding, severe coagulation disorders), psychiatric disorder, or social circumstances that may interfere with trial conduct, compliance, or pose high risk per investigator's judgment.
* Concurrent malignancy diagnosed within <5 years prior to screening.
* Pregnant or lactating women.
* Positive serology for HIV antibody, HBsAg, HCV antibody, or TP antibody at screening.
* Active or latent tuberculosis at screening (positive TB-IGRA test).
* Any other condition deemed ineligible by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 2 years
  A Dose-Limiting Toxicity (DLT) is defined as any adverse event occurring within the 29-day period following the initiation of CC312 intravenous infusion during the dose-escalation phase, assessed by the investigator as related to CC312 and meeting the following criteria: (1) Hematologic Toxicity: Grade 4 toxicity (excluding lymphopenia) persisting beyond 29 days and not attributable to underlying disease; (2) Non-Hematologic Toxicity: Any ≥Grade 4 toxicity potentially related to CC312 during the observation window, or any Grade 3 toxicity potentially related to CC312 that fails to resolve to ≤Grade 2 within 7 days.
Adverse events (AE)/serious adverse events (SAE) | 2 years
  With the exception of CRS and ICANS, which will be graded according to the ASTCT criteria, the severity of all other adverse events (AEs) will be assessed and classified using the CTCAE (Common Terminology Criteria for Adverse Events) version 5.0.

SECONDARY OUTCOMES:
Serum Concentration of CC312 | 2 years
  All subjects are required to undergo blood sampling for serum concentration analysis at the following time points: within 1 hour (0 h) before and 1 hour after the infusion of the priming dose; within 1 hour (0 h) before and 1 hour after the infusion of the first and second doses in weeks 1 and 3, and the first dose in weeks 2 and 4 of the treatment phase; and at early termination or end of study (EOS).
Counts of peripheral B cells | 2 years
  All subjects are required to undergo blood sampling for lymphocyte subset analysis at the following time points: within 1 hour (0 h) before infusion, 1 hour and 24 hours after infusion of the priming dose; within 1 hour (0 h) before infusion, 1 hour and 24 hours after infusion of the first and second doses in weeks 1 and 3 of the treatment phase; within 1 hour (0 h) before the first dose in weeks 2 and 4; during extended dosing after Day 28 (if applicable): within 1 hour before the second weekly dose until the end of the extended dosing period; monthly for 4 consecutive months after the last dose; every 3 months during the long-term follow-up phase; and at early termination or end of study (EOS).
Cytokines | 2 years
  All subjects are required to undergo blood sampling for cytokine analysis (IFN-γ、IFN-α、IL-2、IL-6、IL-10、TNF-α) at the following time points: within 1 hour (0 h) before infusion, 1 hour and 24 hours after infusion of the priming dose during the priming phase; within 1 hour (0 h) before infusion, 1 hour and 24 hours after infusion of the first and second doses in weeks 1 and 3 of the treatment dose phase; within 1 hour (0 h) before infusion, 1 hour and 24 hours after infusion of the first dose in weeks 2 and 4 of the treatment dose phase; and at early termination or end of study (EOS).
Complement | 2 years
  All subjects are required to undergo blood sampling for complement analysis (complements C3 and C4) at the following time points: screening/baseline; within 1 hour (0 h) prior to the priming dose administration; within 1 hour (0 h) prior to the first weekly dose during weeks 1, 2, 3, and 4 of the treatment phase; and at weeks 8, 12, 24, and 48; as well as upon early termination.
Autoantibody | 2 years
  Autoantibody (antinuclear antibody, anti-double stranded DNA antibody, anti-Smith antibody, and antiphospholipid antibody) testing is required at the following time points: within 1 hour (0 h) prior to the priming dose administration, within 1 hour (0 h) prior to the first treatment dose at week 3, and at Day 28; additional autoantibody assessments will be performed at: within 1 hour (0 h) prior to the priming dose, Day 28, Weeks 8, 12, 24, and 48, and upon early termination, with blood samples collected for analysis.
Immunogenicity | 2 years
  All subjects are required to undergo blood sampling for immunogenicity (anti-CC312 antibody) analysis at the following time points: within 1 hour (0 h) prior to the priming dose administration; within 1 hour (0 h) prior to the first weekly dose during weeks 1, 2, 3, and 4 of the treatment phase; and at weeks 8, 12, 16, and 24; as well as upon early termination or end of study (EOS). Blood samples shall be collected at the above-specified time points, with backup aliquots retained, and the actual sampling time recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Deyang People's Hospital, Deyang, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doria A, Amoura Z, Cervera R, Khamastha MA, Schneider M, Richter J, Guillemin F, Kobelt G, Maurel F, Garofano A, Perna A, Murray M, Schmitt C, Boucot I. Annual direct medical cost of active systemic lupus erythematosus in five European countries. Ann Rheum Dis. 2014 Jan;73(1):154-60. doi: 10.1136/annrheumdis-2012-202443. Epub 2012 Dec 21. PMID 23264339
- [Background] Conrad N, Misra S, Verbakel JY, Verbeke G, Molenberghs G, Taylor PN, Mason J, Sattar N, McMurray JJV, McInnes IB, Khunti K, Cambridge G. Incidence, prevalence, and co-occurrence of autoimmune disorders over time and by age, sex, and socioeconomic status: a population-based cohort study of 22 million individuals in the UK. Lancet. 2023 Jun 3;401(10391):1878-1890. doi: 10.1016/S0140-6736(23)00457-9. Epub 2023 May 5. PMID 37156255
- [Background] Karagianni P, Tzioufas AG. Epigenetic perspectives on systemic autoimmune disease. J Autoimmun. 2019 Nov;104:102315. doi: 10.1016/j.jaut.2019.102315. Epub 2019 Aug 15. PMID 31421964